CLINICAL TRIAL: NCT00978419
Title: Randomized, Placebo Controlled, Pilot Trial of Statin Use in Burn Patients
Brief Title: Pilot Trial of Statin Use in Burn Patients
Acronym: BURNSTAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 091060
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-04

CONDITIONS: Burns
Keywords: Statins; Burns; Sedatives; Neurocognitive; Septic; Mortality; C Reactive Protein; Septic shock; Sedation; Neurocognitive function
MeSH Terms: conditions — Burns; Shock, Septic | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin (Active Comparator): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Loading dose 40mg by mouth first day, then 20 mg by mouth for up to 27 days
  Arms: Rosuvastatin
Drug: Placebo — Placebo administered every day for up to 28 days
  Arms: Placebo

SUMMARY:
This is a 90 day study, with patients receiving either oral Rosuvastatin or placebo for up to 28 days. The study will assess the affect of statins administered soon after burn injury on C-reactive protein (CRP) levels, patient mortality and the incidence of septic shock. The investigators also seek to describe the correlation between exposure to statins and development of delirium and de-novo long-term cognitive impairment.

Hypothesis:

1. Statin administration within 96 hours of burn is safe, will decrease CRP, and will decrease septic shock and mortality in burn patients.
2. The investigators hypothesize that burn patients will have a de-novo long term cognitive impairment at 3 months after burn.
3. The investigators hypothesize the use of statins in burn patients will reduce the development and the degree of cognitive impairment at 3 months post burn.

DETAILED DESCRIPTION:
Infection and sepsis are the major causes of morbidity and mortality in burn patients. Several observational studies have shown that HMG-CoA reductase inhibitors, known as statins, before or after illness or injury results in decreased mortality and incidence of sepsis.

We performed a pilot retrospective chart review of 223 patients admitted to the Vanderbilt University Burn Service from 2006-2008 who were ≥55 years of age. Patients were identified as using statin drugs prior to burn, and compared to those who were not. There was a significant decrease in mortality of 83% (P=.004) in the statin group and a 50% reduction in septic shock (p=.155) that was not significant likely due to the low numbers of patients with septic shock (n=30). These effects were unchanged after controlling for cardiovascular comorbidities.

Animal studies have also shown decreased mortality and sepsis with pre-injury statin administration. Mechanisms of statin effect on mortality and septic shock are attributed to the so-called pleiotropic effects.

If the use of statins is potentially expected to reduce mortality, it is even more relevant to understand the long-term cognitive and functional outcomes of the survivors. In the last years researchers highlighted how survivors from acute respiratory distress syndrome (ARDS) largely experience cognitive and functional decline after their acute illness. More recently Jackson et al. advocated a relationship between delirium in intensive care unit (ICU) patients and cognitive impairment; more specifically 1 of 3 survivors of critically illness with delirium developed cognitive impairment. Though every year several patients are admitted to burn units in the United States, to date only one small report has been published addressing the long-term cognitive outcomes of burn ICU patients. In these preliminary data, Varney et al. found that of the eight patients all were found to have significant problems as evidenced in neuropsychological tests, activities of daily living, and from relatives' reports.

The causes of development of a de-novo cognitive impairment in this population are probably multifactorial and could be linked to the development of and duration of delirium or to the exposure to large amount of sedatives-analgesics used to assure the comfort of the patients on the ventilator and to control pain secondary to the burn. ICU delirium is a common acute brain dysfunction with a prevalence as high as 80% in critically ill surgical and medical ICU patients depending on the severity of illness and the instrument used to diagnose delirium. Different risk factors have been called to cause delirium including exposure to drugs. In particular, previous studies have shown how exposure to benzodiazepines (i.e. lorazepam and midazolam) and opiates have been associated to transition to delirium in medical and surgical ICU patients. If sedatives and analgesics are widely used in the medical and surgical ICUs, this is even more striking for the burn units where large amounts of drugs are infused for patient comfort and pain control. Therefore a large exposure to these drugs in burn patients has the potential to influence the prevalence of delirium even more.

Creatine kinase (CK) levels are known to be increased in the serum of burn patients. C-Reactive Protein (CRP) is an hepatically derived acute phase reactant, elevated in burn patients within the first 3 days, and decreases over time. Statins are known to decrease CRP and possibly mitigate the inflammatory response due to CRP.

Rosuvastatin (Crestor) was chosen as the study drug over others for pharmacokinetic and side effect profile.

1. Rosuvastatin has an elimination half-life of 19 hours, making it suitable for once a day dosing.
2. Rosuvastatin is excreted 90% unchanged in the stool, and the other 10% by the liver. (Rosuvastatin drug information, package insert).
3. Rosuvastatin, a hydrophilic statin, seems to be associated with fewer side effects than lipophilic statins and has fewer drug-drug interactions.

Rosuvastatin dose will be 40 mg loading dose first day, then 20mg by mouth or feeding tube daily.

Patients with thermal burn will be recruited on admission to the Vanderbilt University Burn Service within 96 hours from the time of the burn.

The trial will accrue 40 patients admitted to the Burn Service.

Sample size calculation:

alpha = 0.05 power = .80 delta= 200-(.64 * 200) =72(expected difference statin and non-statin subjects) sigma = 80 (95% CI CRP burn patients at 3 days) m = 1 (ratio controls/experimental) Sample size=20

Informed consent will be obtained from the patient or surrogate prior to enrollment in the trial. No study procedures will be done without first obtaining informed consent.

After informed consent is obtained, patients will be assigned to Rosuvastatin or placebo group on a random 1:1 basis. The study will be double blind, with neither the participant, research staff nor clinical staff having knowledge of the treatment assignment until after the database has been locked. Assignment will be made by computer-generated randomization. Placebo will be an inactive tablet provided by the Vanderbilt Investigational Pharmacy that is not distinguishable in appearance from Rosuvastatin.

Patients will be considered to have completed the administration of the study drug when any of the following conditions is met:

1. 28 days after randomization
2. Discharge from the hospital
3. Death

Because CPK is routinely elevated in burn patients and myopathy from statins is very rare and is a delayed side effect, CKs before day 7 of treatment will not be used to trigger the rule for withholding/discontinuing study drug. Values greater than 10 times normal obtained after day 7 will trigger cessation of study drug. Study drug will also be discontinued if the patient develops ALT > 8 times upper limit of normal after study day 1, or if the patient begins treatment with niacin, fenofibrate, cyclosporine, gemfibrozil, lopinavir, ritonavir or oral contraceptives. Data collection will continue as though therapy continued through study day 90.

1. Demographic data (age, sex, race)
2. Medical history, including cardiovascular comorbidities MI, CVA, arrhythmia, PVD, CHF, HTN, DM, COPD
3. Time of burn injury
4. Time of admission to the Burn Service
5. Injury type: burn only, burn plus smoke inhalation
6. Mechanism of burn

   1. structure fire
   2. trauma (i.e., MVA)
   3. scald/steam
   4. grease
   5. contact
   6. home oxygen
   7. flammable liquid
   8. cooking fire
   9. brush fire
   10. other (describe)
7. Extent of burn (% of BSA involved)
8. Physical assessment
9. Sedative drugs during admission, data collected daily.
10. Ventilator days.
11. Activities of Daily Living (ADLs), Instrumental activities of daily living (IADLs)
12. Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE)

Baseline (Day 0) Assessments

The following information will be recorded prior to dosing. If more than one value is available, the closest value prior to the time of dosing will be recorded: serum creatinine, bilirubin, glucose, CK, CRP, PT/PTT/INR and pre-albumin.

4.14 Follow-up Assessments

The following lab results will be recorded at the following timepoints:

1. Serum CK will be collected on days 3, 7, 14, 21, 28.
2. Serum ALT will be collected days 1, 7, 14, 21, 28.
3. Serum CRP will be collected on days 3, 7, 14.

RASS scoring will be assessed and documented at 0800 each day +/- 8 hours. (Appendix B)

Delirium will be evaluated daily with the Confusion Assessment Method in the ICU (CAM- ICU) up to 28 days. (Appendix C)

Type and total amount of sedatives and analgesic drugs will be collected daily up to 28 days.

The ADL 41 and the Mini Mental State Examination (MMSE) will be evaluated at hospital discharge. (Appendix D)

At a 3-month follow-up patients will be evaluated with the ADL, IADL, MMSE, Hospital Anxiety and Depression Scale (HADS), and the EuroQol.(Appendix E, F, G) The use of analgesics will also be collected.

Data will be analyzed using STATA 9 statistical program. Demographics, characteristics of burn, primary and secondary endpoints will be tabulated and compared across Rosuvastatin and placebo groups. CRP levels by Rosuvastatin use and occurrence of septic shock will be analyzed using area under the curve (AUC). Mortality and occurrence of septic shock adjusted for cardiovascular co-morbidities will be examined using multivariate logistic regression.

Potential risks of study drug include:

1. Myopathy, defined as CK > 10 times ULN, which has been reported in < .01% of patients, is usually reversible with discontinuation of the statin. Rhabdomyolysis, severe myopathy, defined as CK > 40 times ULN, can be expected in about a third of those, can lead to renal failure from myoglobin release, requires stopping the study drug, hydration and medical treatment.
2. Increase in liver enzymes (in our study ALT > 8 times ULN) after day 1, reported in .08% after 4 months of statin use, and drug interactions. Simple discontinuation of the drug is sufficient as there is no evidence that liver failure will ensue.23
3. Additional uncommon risks of study drug include: headache, nausea, myalgia, asthenia, abdominal pain, dizziness, and constipation, from the package insert.

We will monitor CK and ALT levels and discontinue study drug if defined toxicity levels are reached. CK and ALT levels that meet toxicity levels will be reported as adverse events. Myopathy will be noted as an adverse event, but will not by itself stop study drug unless associated with CK levels as defined.

Adverse Event Recording Each adverse event occurring to a subject / patient, either spontaneously revealed by the patient / subject or observed by the Investigator, whether believed by the Investigator to be related or unrelated to the study drug, must be recorded on the adverse event information page of the CRF and on the patient / subject's hospital/center notes.

The Investigator will also determine the relationship of any adverse event to study drug and record it on the appropriate section of the CRF as well as their intensity, time of onset, duration, and the precautions carried out. The Investigator must record all adverse events, which occur during the study, regardless of their relationship to study drug and if they occur during a period without administration of study medication.

Adverse Event Reporting Investigators will assess the subject and medical record to determine if adverse experiences occur during the 60 day study or to hospital discharge, whichever occurs first. The investigator will determine if any changes in laboratory values or clinical signs are those expected in the course of a patient with burn injuries.

Always reported as adverse events:

CK> 10 times ULN after study day 7 ALT> 8 times ULN after study day 1

Serious Adverse Events will have to be reported according to the following special procedure:

The Investigator will report SAE's to the Vanderbilt Institutional Review Board per policy. All serious adverse events that occur in association with the study will be reviewed by study personnel and reported to the Vanderbilt Institutional Review Board (IRB) within 10 days of the Investigator's awareness of the event. Any new information that comes to light which may affect the subject or their caregiver's decision to continue to participate in the study will be passed on to them as soon as possible. This may also result in a change to the consent form and review by the IRB. Serious adverse events will also be reported to and reviewed by the data safety monitor.

8.0 Privacy/Confidentiality Issues

The Principal investigator will collect data and enter it into password protected computer in a locked office. Each patient will have a unique identifier number, with the key to the patient's medical record number kept in a locked cabinet in the office. Only research associates or those individuals directly involved with the study will have access to data. Information is for research purposes only and when used for publication purposes, all participants will have their names concealed. Access to identified patient information will be limited to the investigators listed within the IRB application. De-identified information with HIPAA identifiers removed will be available to other investigators following IRB approval. Confidentiality and security will be maintained for the database. The database is stored behind a firewall (in addition to the institutional firewall) with the highest level of protection, i.e. the same level of protection as the on-line hospital information system at Vanderbilt. This means that users must logon to a web server that sits between the institutional firewall and the firewall to the database, and only this application server is allowed to query the database. Only users approved through our institutional review board will be allowed access to patient identifiers. Other levels of authorization may exist for future approved users following IRB approval, e.g. access to de-identified data.

Data is initially collected in the medical record for each individual study participant. The information will be extracted from the patient's medical record and then transferred into the Case Report Form (CRF). The study data will be kept on site and in a securely locked room to protect patient confidentiality.

The CRFs do not include personal identifiers for any participant. Numbers and initials are assigned for each participant and these become the identifying information for each study participant. A master list is kept separately that identifies which names go with which numbers and initials.

Study personnel (PI and co-investigators) and government regulatory agencies have access to all research records as required by law. Others (such as law enforcement agencies) may have access to records as defined by law.

Follow-up and Record Retention

The study records will be stored for investigation for at least six years and may be retained indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Thermal burn occurring within the 96 hours prior to dosing

Exclusion Criteria:

* Inability to obtain informed consent (or assent from surrogate)
* Less than 18 years of age
* Patient or surrogate not committed and/or not likely to remain committed to full support, as, for example, would be the case for a patient with end-stage cancer or other end-stage terminal conditions. Commitment to full support need not include cardiopulmonary resuscitation provided the team is committed to other forms of full support
* Unable to receive or absorb enteral study drug
* Statin specific exclusions
* Receiving a statin medication within 48 hours of dosing (to exclude controls from exposure to statins)
* Allergy or intolerance to statins
* ALT or AST > 5 times upper limit of normal
* Untreated hypothyroidism by history (package insert)
* Pregnancy or breastfeeding
* Receiving niacin, fenofibrate, cyclosporine, gemfibrozil, lopinavir, ritonavir or oral contraceptives within 24 hours prior to admission (package insert)
* Advanced cirrhosis, defined as a history of chronic liver disease and a Child-Pugh Class score >10 (Appendix A)
* Moribund patient not expected to survive 24 hours
* Patients admitted to the Burn Service for non-thermal burn conditions, including chemical burn, TENS, electrical injury or wound care
* Patient expected to be discharged within 24 hours
* Patients of Asian descent (due to pharmacokinetics issues with Rosuvastatin in this population)
* Patients receiving another interventional investigational drug within the 30 days prior to dosing
* Patients otherwise unsuitable for participation in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Bloemsma GC, Dokter J, Boxma H, Oen IM. Mortality and causes of death in a burn centre. Burns. 2008 Dec;34(8):1103-7. doi: 10.1016/j.burns.2008.02.010. Epub 2008 Jun 6. PMID 18538932
- [Background] Woodward B, Cartwright M. Safety of drotrecogin alfa (activated) in severe sepsis: data from adult clinical trials and observational studies. J Crit Care. 2009 Dec;24(4):595-602. doi: 10.1016/j.jcrc.2008.11.011. Epub 2009 Feb 12. PMID 19327331
- [Background] Almog Y, Shefer A, Novack V, Maimon N, Barski L, Eizinger M, Friger M, Zeller L, Danon A. Prior statin therapy is associated with a decreased rate of severe sepsis. Circulation. 2004 Aug 17;110(7):880-5. doi: 10.1161/01.CIR.0000138932.17956.F1. Epub 2004 Aug 2. PMID 15289367
- [Background] Chua D, Tsang RS, Kuo IF. The role of statin therapy in sepsis. Ann Pharmacother. 2007 Apr;41(4):647-52. doi: 10.1345/aph.1H550. Epub 2007 Mar 27. PMID 17389664
- [Background] Merx MW, Weber C. Statins in the intensive care unit. Curr Opin Crit Care. 2006 Aug;12(4):309-14. doi: 10.1097/01.ccx.0000235207.00322.96. PMID 16810040
- [Background] Efron DT, Sorock G, Haut ER, Chang D, Schneider E, Mackenzie E, Cornwell EE 3rd, Jurkovich GJ. Preinjury statin use is associated with improved in-hospital survival in elderly trauma patients. J Trauma. 2008 Jan;64(1):66-73; discussion 73-4. doi: 10.1097/TA.0b013e31815b842a. PMID 18188101
- [Background] Fogerty MD, Efron D, Morandi A, Guy JS, Abumrad NN, Barbul A. Effect of preinjury statin use on mortality and septic shock in elderly burn patients. J Trauma. 2010 Jul;69(1):99-103. doi: 10.1097/TA.0b013e3181df61b1. PMID 20622585
- [Background] Merx MW, Liehn EA, Graf J, van de Sandt A, Schaltenbrand M, Schrader J, Hanrath P, Weber C. Statin treatment after onset of sepsis in a murine model improves survival. Circulation. 2005 Jul 5;112(1):117-24. doi: 10.1161/CIRCULATIONAHA.104.502195. PMID 15998696
- [Background] Merx MW, Liehn EA, Janssens U, Lutticken R, Schrader J, Hanrath P, Weber C. HMG-CoA reductase inhibitor simvastatin profoundly improves survival in a murine model of sepsis. Circulation. 2004 Jun 1;109(21):2560-5. doi: 10.1161/01.CIR.0000129774.09737.5B. Epub 2004 May 3. PMID 15123521
- [Background] Lennernas H, Fager G. Pharmacodynamics and pharmacokinetics of the HMG-CoA reductase inhibitors. Similarities and differences. Clin Pharmacokinet. 1997 May;32(5):403-25. doi: 10.2165/00003088-199732050-00005. PMID 9160173
- [Background] Istvan ES, Deisenhofer J. Structural mechanism for statin inhibition of HMG-CoA reductase. Science. 2001 May 11;292(5519):1160-4. doi: 10.1126/science.1059344. PMID 11349148
- [Background] Terblanche M, Almog Y, Rosenson RS, Smith TS, Hackam DG. Statins and sepsis: multiple modifications at multiple levels. Lancet Infect Dis. 2007 May;7(5):358-68. doi: 10.1016/S1473-3099(07)70111-1. PMID 17448939
- [Background] Gao F, Linhartova L, Johnston AM, Thickett DR. Statins and sepsis. Br J Anaesth. 2008 Mar;100(3):288-98. doi: 10.1093/bja/aem406. PMID 18276651
- [Background] Imaki M, Miyoshi T, Tanada S, Nakamura T, Yamada Y, Yamasaki R, Terada H. Effect of lard and corn oil intake on serum lipids in young men. Acta Biol Hung. 1989;40(3):271-82. PMID 2633589
- [Background] McGown CC, Brookes ZL. Beneficial effects of statins on the microcirculation during sepsis: the role of nitric oxide. Br J Anaesth. 2007 Feb;98(2):163-75. doi: 10.1093/bja/ael358. PMID 17251210
- [Background] Hopkins RO, Weaver LK, Chan KJ, Orme JF Jr. Quality of life, emotional, and cognitive function following acute respiratory distress syndrome. J Int Neuropsychol Soc. 2004 Nov;10(7):1005-17. doi: 10.1017/s135561770410711x. PMID 15803563
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Varney NR, Ju D, Shepherd JS, Kealey GP. Long-term neuropsychological sequelae of severe burns. Arch Clin Neuropsychol. 1998 Nov;13(8):737-49. PMID 14590632
- [Background] McNicoll L, Pisani MA, Zhang Y, Ely EW, Siegel MD, Inouye SK. Delirium in the intensive care unit: occurrence and clinical course in older patients. J Am Geriatr Soc. 2003 May;51(5):591-8. doi: 10.1034/j.1600-0579.2003.00201.x. PMID 12752832
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Peterson JF, Pun BT, Dittus RS, Thomason JW, Jackson JC, Shintani AK, Ely EW. Delirium and its motoric subtypes: a study of 614 critically ill patients. J Am Geriatr Soc. 2006 Mar;54(3):479-84. doi: 10.1111/j.1532-5415.2005.00621.x. PMID 16551316
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Costabile S, Truman Pun B, Dittus R, Ely EW. Motoric subtypes of delirium in mechanically ventilated surgical and trauma intensive care unit patients. Intensive Care Med. 2007 Oct;33(10):1726-31. doi: 10.1007/s00134-007-0687-y. Epub 2007 Jun 5. PMID 17549455
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Dubois MJ, Bergeron N, Dumont M, Dial S, Skrobik Y. Delirium in an intensive care unit: a study of risk factors. Intensive Care Med. 2001 Aug;27(8):1297-304. doi: 10.1007/s001340101017. PMID 11511942
- [Background] Pandharipande P, Shintani A, Peterson J, Pun BT, Wilkinson GR, Dittus RS, Bernard GR, Ely EW. Lorazepam is an independent risk factor for transitioning to delirium in intensive care unit patients. Anesthesiology. 2006 Jan;104(1):21-6. doi: 10.1097/00000542-200601000-00005. PMID 16394685
- [Background] Pandharipande P, Cotton BA, Shintani A, Thompson J, Pun BT, Morris JA Jr, Dittus R, Ely EW. Prevalence and risk factors for development of delirium in surgical and trauma intensive care unit patients. J Trauma. 2008 Jul;65(1):34-41. doi: 10.1097/TA.0b013e31814b2c4d. PMID 18580517
- [Background] Brown C, Albrecht R, Pettit H, McFadden T, Schermer C. Opioid and benzodiazepine withdrawal syndrome in adult burn patients. Am Surg. 2000 Apr;66(4):367-70; discussion 370-1. PMID 10776874
- [Background] Guechot J, Lioret N, Cynober L, Letort C, Saizy R, Giboudeau J. Myoglobinemia after burn injury: relationship to creatine kinase activity in serum. Clin Chem. 1986 May;32(5):857-9. PMID 3698276
- [Background] Barati M, Alinejad F, Bahar MA, Tabrisi MS, Shamshiri AR, Bodouhi NO, Karimi H. Comparison of WBC, ESR, CRP and PCT serum levels in septic and non-septic burn cases. Burns. 2008 Sep;34(6):770-4. doi: 10.1016/j.burns.2008.01.014. Epub 2008 May 29. PMID 18513877
- [Background] Dehne MG, Sablotzki A, Hoffmann A, Muhling J, Dietrich FE, Hempelmann G. Alterations of acute phase reaction and cytokine production in patients following severe burn injury. Burns. 2002 Sep;28(6):535-42. doi: 10.1016/s0305-4179(02)00050-5. PMID 12220910
- [Background] Ulrich D, Noah EM, Pallua N. [Plasma endotoxin, procalcitonin, C-reactive protein, and organ functions in patients with major burns]. Handchir Mikrochir Plast Chir. 2001 Jul;33(4):262-6. doi: 10.1055/s-2001-16595. German. PMID 11518988
- [Background] Aguilar EM, Miralles Jde H, Gonzalez AF, Casariego CV, Moreno SB, Garcia FA. In vivo confirmation of the role of statins in reducing nitric oxide and C-reactive protein levels in peripheral arterial disease. Eur J Vasc Endovasc Surg. 2009 Apr;37(4):443-7. doi: 10.1016/j.ejvs.2008.12.009. Epub 2009 Feb 10. PMID 19211277
- [Background] Irimura T, Nakajima M, Hirano H, Osawa T. Distribution of ferritin-conjugated lectins on sialidase-treated membranes of human erythrocytes. Biochim Biophys Acta. 1975 Dec 1;413(2):192-201. doi: 10.1016/0005-2736(75)90103-0. PMID 172150
- [Background] Doggrell SA. Relating statin therapy to C-reactive protein levels. Expert Opin Pharmacother. 2005 Aug;6(9):1597-600. doi: 10.1517/14656566.6.9.1597. PMID 16086647
- [Background] Armitage J. The safety of statins in clinical practice. Lancet. 2007 Nov 24;370(9601):1781-90. doi: 10.1016/S0140-6736(07)60716-8. PMID 17559928
- [Background] Sachse C, Machens HG, Felmerer G, Berger A, Henkel E. Procalcitonin as a marker for the early diagnosis of severe infection after thermal injury. J Burn Care Rehabil. 1999 Sep-Oct;20(5):354-60. doi: 10.1097/00004630-199909000-00004. PMID 10501320
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Pfeffer RI, Kurosaki TT, Harrah CH Jr, Chance JM, Filos S. Measurement of functional activities in older adults in the community. J Gerontol. 1982 May;37(3):323-9. doi: 10.1093/geronj/37.3.323. PMID 7069156
- [Background] Jorm AF, Jacomb PA. The Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE): socio-demographic correlates, reliability, validity and some norms. Psychol Med. 1989 Nov;19(4):1015-22. doi: 10.1017/s0033291700005742. PMID 2594878
- [Background] Jorm AF, Scott R, Cullen JS, MacKinnon AJ. Performance of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) as a screening test for dementia. Psychol Med. 1991 Aug;21(3):785-90. doi: 10.1017/s0033291700022418. PMID 1946866
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Levy MM, Fink MP, Marshall JC, Abraham E, Angus D, Cook D, Cohen J, Opal SM, Vincent JL, Ramsay G; SCCM/ESICM/ACCP/ATS/SIS. 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference. Crit Care Med. 2003 Apr;31(4):1250-6. doi: 10.1097/01.CCM.0000050454.01978.3B. PMID 12682500

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Both Principal Investigators left Vanderbilt without completing record. Have been unable to find any records from this study or publication. Total enrollment and completion date are from IRB records.
Period: Overall Study
Arm/Group | Rosuvastatin | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Reduction in CRP Level Over Time, Compared to Placebo Measured at Baseline and Days 3, 7, 14. The Mean CRP Levels at Specified Days Will be the Endpoints.
Time Frame: Days 1, 3, 7, 14
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mortality Compared to Placebo
Time Frame: 90 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mortality Compared to Placebo, Adjusted for Cardiovascular Co-morbidities
Time Frame: 90 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Reduction in the Incidence of Septic Shock (See Definition) Compared to Placebo
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Reduction in the Incidence of Septic Shock (See Definition) Compared to Placebo, Adjusted for Cardiovascular Co-morbidities
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: A Reduction in CK Levels Over Time, Compared to Placebo Measured at Baseline and Days 3, 7, 14, 21, 28
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: A Reduction in ALT Levels Over Time, Compared to Placebo, Measured at Baseline, Days 1, 7, 14, 21, 28
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Determine the Safety of Rosuvastatin Compared to Placebo in Burn Patients by Comparing the Frequency, Type and Severity of Adverse Events
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Determine Which Are Appropriate Attainable Endpoints for Future Trials and the Number of Participants Required to Reach Significance in Analysis of a Variety of Variables
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Determine the Prevalence of Delirium in the Two Subgroup of Patients
Time Frame: 28 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Determine the Prevalence of De-novo Long-term Neurocognitive Impairment in Burn Patients and by Study Group.
Time Frame: 90 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Determine the Prevalence of Functional Impairment in Burn Patients and by Study Group
Time Frame: 90 days
Arm/Group | Rosuvastatin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Rosuvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes